CLINICAL TRIAL: NCT03743922
Title: The Effects of Vitamin D2 Supplement During Pregnancy on Postpartum Maternal and Fetal Vitamin D Levels: the Randomized Controlled Trial
Brief Title: The Effects of Vitamin D2 Supplement During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THAIVITD2
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy Early
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral calciferol group (Experimental): Subjects will receive oral calciferol 20,000 iu per week during pregnancy until delivered
  Interventions: Drug: Calciferol
- oral placebo group (Placebo Comparator): Subjects will receive oral placebo 1 tab per week during pregnancy until delivered
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calciferol — calciferol capsule
  Other Names: vitimin d2
  Arms: Oral calciferol group
Drug: Placebo — placebo capsule
  Other Names: placebo ( for calciferol )
  Arms: oral placebo group

SUMMARY:
The effects of vitamin D2 supplement during pregnancy on postpartum maternal and fetal vitamin D levels: the randomized controlled trial

DETAILED DESCRIPTION:
Vitamin D structurally similar to steroids. Made from the skin. And metabolism of the liver, kidneys, vitamin D levels in the bloodstream are two types of vitamin D 2 (Ergocalciferol) and vitamin D 3 (Cholecalciferol) Vitamin D regulates calcium and phosphorus levels in the body. Including the accumulation of minerals in the bone. Vitamin D is important in the formation of bones and teeth and the normal growth of children, affects the reabsorption of amino acids in the kidneys, regulates the amount of calcium and phosphorus in the blood Vitamin D deficiency in pregnant affects the mother and baby example high maternal blood pressure during pregnancy, diabetes during pregnancy, increase birth body weight of baby. low calcium seizures Infants, baby have bones and growth disorders. Currently, no vitamin D supplement is used in pregnant women in Thailand who attend antenatal clinics. The researcher has proposed to study the effects of vitamin D supplement during pregnancy on postpartum maternal and fetal vitamin D levels by using vitamin D 20,000IU / week

ELIGIBILITY:
Inclusion Criteria:

* Women who have pregnant and ANC at Rajavithi hospital
* Women who have age at least 18 year
* Women who have Thai nationality
* Women who have pregnant of gestational age under 20week

Exclusion Criteria:

* Women who don't plan of delivered at Rajavithi hospital
* Women who have complication of pregnancy
* Woman who delivered before gestational age 37week
* Women who have abnormal kidney function
* Woman who have been used anticonvulsant drug or others form of vitamin d
* Women who have vitamin d allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
effect of vitamin D 2 supplementation during pregnancy | within 30 minute after delivered
  To study the effect of vitamin D 2 supplementation during pregnancy on postpartum maternal and fetal vitamin D levels effects of vitamin D2 supplement during pregnancy on postpartum maternal and fetal vitamin D levels

SECONDARY OUTCOMES:
vitamin D levels in maternal blood during pregnancy | at first time ANC
  To assess vitamin D levels in maternal blood during pregnancy
vitamin D levels in maternal blood after vitamin D supplementation | within 30 minute after delivered
  To assess vitamin D levels in maternal blood after vitamin D supplementation during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Patitta Vacharaprechaskul, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi hospital, Bangkok, Thailand, Thailand

IPD SHARING:
Plan to Share IPD: Undecided